CLINICAL TRIAL: NCT02895581
Title: Retrospective Study of the Survival of Patients Suffering From Hiv-related Progressive Multifocal Leukoencephalopathy
Acronym: LEMPMAR
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_AMR_2015_1
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Progressive Multifocal Leukoencephalopathy
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Retrospective medical chart review of HIV-infected patients diagnosed with progressive multifocal leukoencephalopathy

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients
* Diagnosed with progressive multifocal leukoencephalopathy
* Minimal follow-up of one year OR patient deceased less than one year after diagnosis

Exclusion Criteria:

* Loss of follow-up within 12 months after diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients diagnosed with progressive multifocal leukoencephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2006-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Rankin score | 12 months after diagnosis of leukoencephalopathy